CLINICAL TRIAL: NCT06026176
Title: Pattern of Clinical Presentation of Different Breast Disease in Surgical Opd at BPKIHS
Status: Completed | Type: Observational
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Sishir Poudel, Doctor, B.P. Koirala Institute of Health Sciences
Other Study IDs: IRC/2433/022
Record Dates: First submitted 2023-08-18; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Breast Disease; Breast Neoplasms; Breast Pain; Breast Fibroadenoma
MeSH Terms: conditions — Breast Diseases; Breast Neoplasms; Mastodynia; Fibroadenoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Research Title PATTERN OF CLINICAL PRESENTATION OF DIFFERENT BREAST DISEASE IN SURGICAL OPD AT BPKIHS

Rationale: The Study will help us to know about pattern of presentation of different breast diseases

Aims and Objectives:

1. To investigate the pattern of symptoms in patients with Breast diseases
2. To assess the burden of different Breast diseases. Research Hypothesis (if relevant): N/A

1. Material & Methods:

1. Whether study involves Human/animals or both : Human
2. Population/ participants: Files of patients presenting in Surgical OPD with Breast related complaints
3. Type of study design: : Descriptive Research Design
4. Human study :

   Inclusion Criteria: Patients presenting in Surgical OPD with Breast and related complaints Exclusion Criteria: Those who deny consent for participation.
5. Expected sample size : 823 Sample size calculation: Mentioned in methodology
6. Control groups : N/A
7. Probable duration of study: 365 days
8. Setting: Outpatient Department
9. Parameter/Variables to be applied/measured Independent Variables i. Socio-demographic characteristics such as age, gender, address. ii. Family History

Dependent Variables:

i. Clinical symptoms associated with breast disease ii. Type of breast disease (benign or malignant)

Outcome measures:

Primary (main outcome): All dependent variables

(i) Rational for statistical methods to be employed : Retrospective Study Data will be entered in Microsoft Excel and converted it into SPSS for statistical analysis For descriptive studies, percentage, ratio, mean, SD, median will be calculated along with graphical and tabular presentations.

For inferential statistics, bivariate analysis will be done using χ2 test and independent t test to find out the significant differences between dependent and independent variables at 95% confidence interval and p-value significant at <0.05. Multivariate logistic regression will be done to adjust for confounding.

(ii) Ethical clearance : Ethical clearance will be obtained from Under Graduate Medical Research Protocol Review Board (UM-RPRB) of BPKIHS.

(iii) Permission to use copyright questionnaire/Pro forma: Not applicable

(j) Maintain the confidentiality of subject Confidentiality of the participants will be maintained. Whether available resources are adequate: Yes

1. Other resources needed: No
2. For Intervention trial: Not applicable A. Permission from Drug Controller of Nepal required/ Not required/Received/ Applied when_____ B. Safety measure C. Plan to withdraw

DETAILED DESCRIPTION:
Pattern of clinical presentation of different breast disease in surgical opd at BPKIHS

INTRODUCTION

Breast is a dynamic gland that experiences physiological changes throughout a female's reproductive years. Adolescence, menarche, and menopause are notable periods during which significant changes occur in the breasts. Breast diseases are more prevalent in females and encompass a spectrum of benign, infectious, and malignant disorders. Benign breast diseases, constituting the majority of cases, encompass a range of lesions, including developmental abnormalities, inflammatory lesions, epithelial, and stromal proliferations, as well as various neoplasms.

Benign breast disease is the primary cause of breast problems, with up to 30% of women experiencing a benign breast disorder that requires treatment at some point in their lives. The most common symptoms associated with these disorders are pain, lumpiness, or the presence of a lump.

Breast cancer is most commonly observed in the Western world and is extremely rare before the age of 20 years. It is also rare in males. Breast cancer occurs more frequently in women with a family history of the disease. The typical presentation of breast cancer involves the presence of a hard lump, which may be associated with indrawing of the nipple or overlying skin.

A study conducted in Nepal revealed that benign breast conditions accounted for 61.7% of cases, while malignancy accounted for 15.3%.

Pain is one of the most common breast symptoms experienced by women. Breast pain is typically classified as cyclical mastalgia, noncyclical mastalgia, or extra mammary (non-breast) pain. Cyclic mastalgia is breast pain that follows a clear relationship to the menstrual cycle. Noncyclic mastalgia may be constant or intermittent and is not linked to the menstrual cycle; it often occurs after menopause. Extramammary pain arises from the chest wall or other sources but is interpreted as originating within the breast. The risk of cancer in a woman presenting with breast pain as her only symptom is extremely low.

Breast lump/mass is also one of the most common breast symptoms. The discovery of a breast mass, whether self-detected or identified by a clinician, is a common and often distressing occurrence for many women. Although most detected breast masses are benign, it is essential for every woman presenting with a breast mass to undergo evaluation to rule out or diagnose cancer.

Nipple discharge ranks as the third most common breast complaint, following breast pain and breast mass. It is usually a benign condition and can present in several forms, including milky, multicolored and sticky, purulent, clear and watery, yellow or serous, pink or serosanguinous, and bloody or sanguinous. The characteristics of the nipple discharge aid in the early diagnosis and management of breast disease. The most common cause of pathologic nipple discharge is a benign papilloma, followed by ductal ectasia, while carcinoma is the least likely cause.

Breast diseases represent a significant health concern worldwide, including Nepal. Despite this, there have been relatively few studies conducted in Nepal to investigate the spectrum of breast diseases, and the available studies have been limited by small sample sizes. The current study aims to address this knowledge gap by examining the demographic profile of breast-related diseases and the rate of malignancy in our specific setting. The findings of this study can provide valuable information for healthcare providers in Nepal to improve early detection and management of breast diseases. Furthermore, it can serve as a foundation for future research to better understand the burden and nature of breast diseases in our population. This study's contribution to the global knowledge of breast diseases is particularly valuable, especially in countries with limited resources and healthcare infrastructure. Ultimately, the study seeks to enhance health outcomes and improve the quality of life for individuals affected by breast diseases in Nepal.

In a study conducted in Olabisi Onabanjo University Teaching Hospital in Nigeria, breast lump was the commonest clinical feature of breast disease. Over 60% of these were benign. Breast pain was a statistically significant presentation in patients with malignant breast disease.

In a study carried out at Chaudhry Rehmat Ali Memorial Trust Teaching Hospital Township Lahore, the commonest presentation was lump breast alone and it accounted for 50 patients of 142(35%). The other common symptom was lumpiness (19%) and pain in breast (14%).

In a prospective study conducted in HBS Hospital Islamabad, which included total of 225 female patients, frequency of the disorders was as follows. Fibroadenoma breast presenting as lump breast was found in n=69(30.6%) followed by cyclical mastalgia(n=62 (27.5%), breast abscess n=27(12%), duct ectasia n=18(8%), carcinoma breast n=13(5.7%), sebaceous cyst breast n=9(4%), mastitis n=8(3%), cracked nipples n=8(3%), noncyclical mastalgia n=4(1.7%), galactorrhea n=3(0.8%), breast budding n=1(0.4%), phyllodes tumor n=1(0.4%), blood stained nipple discharge n=1(0.4%) and nipple eczema n=1(0.4%).

In a three years study done in Maheshwara Medical College and Hospital in India 117 patients (110 Female and 7 Male) were studied. The maximum number of patients presented clinically with a lump in the breast (31.81%) and the second symptom was a pain in the breast (27.37%). The common breast diseases were benign and malignant neoplasms. In the benign conditions, most common was fibroadenoma (69 patients 62.72%) in young females. In older age >40 years, the breast cancer was common. All the seven male patients with breast enlargement clinically, diagnosed as gynecomastia and histopathologically confirmed.

A prospective descriptive study conducted between January 2015 and May 2015 at Manipal Teaching Hospital, a tertiary level hospital situated in western region of Nepal where 160 patients presenting with benign breast diseases were studied. Majority were female (96%). The commonest presentation of benign breast diseases was pain (45%), followed by lump (26%). Fibroadenoma accounted for 46%. This study showed that among the benign breast diseases in females there were preponderance of mastalgia and fibroadenoma followed by fibrocystic diseases.

METHODS

The research utilized a Descriptive Research Design to investigate various study variables. The study focused on socio-demographic characteristics such as age, sex, and address, as well as breast symptoms like pain, lump, discharge, nipple retraction, and sub-areolar fistula. These factors served as outcome variables in the study. The research was conducted at B.P. Koirala Institute of Health Sciences (BPKIHS), and the study population consisted of patients who presented with breast and related complaints in the Surgical OPD. The sampling method included all patients who attended the surgical OPD with breast-related complaints, and data was collected using a semi-structured questionnaire through interviews. The sample size was justified based on literature review and prevalence study calculations. Inclusion criteria were patients who presented in the Surgical OPD with relevant complaints, while those who denied consent were excluded. The data collection involved a validated proforma with sections on sociodemographic profiles and contextual information related to presenting symptoms and family history. Consent was obtained, and English or Nepali questionnaires were used based on participant preference.

Data entry was done in Microsoft Excel and the investigators used SPSS v11.5 for statistical analysis. We used descriptive and inferential statistical methods for data analysis. Descriptive statistics were presented in percentage, ratio, mean, SD and median along with presentation in graphical form. Categorical variables were analyzed with the χ2 test or with Fisher's exact test if at least one cell had an expected count < 5. P value <0.05 was considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting in Surgical OPD with Breast and related complaints

Exclusion Criteria:

* Those who deny consent for participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who presented to the surgical outpatient department (OPD) of a community-based tertiary care hospital in Nepal. These patients sought medical attention for various breast-related complaints over a one-year period. The population includes both male and female individuals.
Sampling Method: Non-Probability Sample
Enrollment: 1023 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Clinical symptoms associated with breast disease | One year
Type of breast disease (benign or malignant) | One Year

CONTACTS AND LOCATIONS:
Locations (1):
- BPKIHS, Dharān, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: Undecided